CLINICAL TRIAL: NCT03557281
Title: A Phase IIa Open-label Trial to Investigate the Early Bactericidal Activity, Safety and Tolerability of GSK3036656 in Participants With Drug-sensitive Pulmonary Tuberculosis
Brief Title: An Early Bactericidal Activity, Safety and Tolerability of GSK3036656 in Subjects With Drug-sensitive Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201214
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Tuberculosis
Keywords: Early bactericidal activity; Mycobacterium Tuberculosis; GSK3036656; Pulmonary tuberculosis; Colony forming units
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — GSK656

STUDY DESIGN:
Intervention Model Description: Eligible subjects in each cohort will be randomized to receive sequential doses of either GSK3036656 or standard-of-care (RIFAFOUR) regimen. This study will employ dose escalation, where the decision to proceed to each subsequent dose level will be made based on safety, tolerability and preliminary pharmacokinetic data from the prior cohort.
Masking Description: This will be an open label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Rifafour e-275 (Active Comparator): All participants will receive a standard-of-care therapy (rifafour e-275) tablet, orally, once daily from Day 1 to Day 14. Participants will receive the standard treatment for tuberculosis (i.e. rifafour e-275 or equivalent generic alternative) once the study treatment (Day 1 to Day 14) is completed.
  Interventions: Drug: Rifafour e-275
- GSK3036656 1 mg (Experimental): Participants will receive a loading dose of GSK3036656 3 milligram (mg), capsule, orally on Day 1, followed by maintenance dose of GSK3036656 1 mg, orally, once daily from Day 2 to Day 14.
  Interventions: Drug: GSK3036656
- GSK3036656 5 mg (Experimental): Participants will receive a loading dose of GSK3036656 15 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 5 mg, orally, once daily from Day 2 to Day 14.
  Interventions: Drug: GSK3036656
- GSK3036656 15 mg (Experimental): Participants will receive a loading dose of GSK3036656 30 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 15 mg, orally, once daily from Day 2 to Day 14.
  Interventions: Drug: GSK3036656
- GSK3036656 30 mg (Experimental): Participants will receive a loading dose of GSK3036656 75 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 30 mg, orally, once daily from Day 2 to Day 14.
  Interventions: Drug: GSK3036656

INTERVENTIONS:
Drug: GSK3036656 — GSK3036656 will be administered
  Arms: GSK3036656 1 mg; GSK3036656 15 mg; GSK3036656 30 mg; GSK3036656 5 mg
Drug: Rifafour e-275 — Rifafour e-275 will be administered
  Arms: Rifafour e-275

SUMMARY:
Tuberculosis remains a concerning health problem, with Mycobacterium Tuberculosis (MTB) now causing more deaths than acquired immune deficiency syndrome (AIDS). GSK3036656 is a compound with a novel mechanism of action under development for the treatment of tuberculosis. It suppresses protein synthesis in MTB by selectively inhibiting the enzyme Leucyl t-ribose nucleic acid (RNA) synthetase. Thus, this study will investigate the early bactericidal activity, safety and tolerability of GSK3036656 in up to four sequential cohorts of subjects with rifampicin-susceptible tuberculosis. The primary objective of this dose-escalation study is to establish the anti-tuberculosis effect of GSK3036656 on serial colony forming units (CFU) counts of MTB in sputum over 14 days of therapy. Subjects in each cohort will be randomized in 3:1 ratio to one of two treatments: either GSK3036656 or standard-of-care (RIFAFOUR® e-275) regimen. The approximate duration of the study for an individual subject will be 5 weeks, including 1 week of screening, 2 weeks of treatment period and another 2 weeks of final follow-up visit. RIFAFOUR e-275 is a registered trademark of Sanofi-Aventis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* In addition, subjects recruited into cohorts that are planned to undergo fluorodeoxyglucose (FDG) positron emission tomography/ Computed Tomography (PET/CT) must be >=25 years of age, at the time of signing the informed consent.
* New episode of untreated, rifampicin-susceptible pulmonary tuberculosis.
* A chest X-ray picture which in the opinion of the Investigator is consistent with tuberculosis.
* At least one sputum sample positive on direct microscopy for acid-fast bacilli (at least 1+ on the International Union Against Tuberculosis and Lung Disease/ World Health Organization [IUATLD/WHO] scale) or molecular test (Xpert MTB/ rifampicin) with result of either medium or high positive for MTB: Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 milliliter or more); estimated from a spot sputum sample at screening; confirmed at the first overnight collection; if less than 10 milliliter is collected overnight this may be repeated once.
* Normal echocardiogram or echocardiogram with normal left ventricular function with at most trace to mild valvular regurgitation and no valvular stenosis.
* Within the normal range for the assay for troponin and b-type natriuretic peptide at screening.
* Body weight (in light clothing and with no shoes) between 40 and 90 kilograms, inclusive, at screening.
* Male or female of non-childbearing potential will be included in the study. A male subject with female partners of child-bearing potential must agree to use contraception during the treatment period and for at least 6 weeks, corresponding to time needed to eliminate study treatment plus an additional 90 days (a spermatogenesis cycle) for study treatments with teratogenic potential after the last dose of study treatment and refrain from donating sperm during this period. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Pre-menopausal females with one of the following; documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or documented bilateral salpingectomy; hysterectomy; documented Bilateral Oophorectomy. Postmenopausal will be defined as 12 months of spontaneous amenorrhea without an alternative medical cause. Post-menopausal status will be confirmed by a simultaneous follicle-stimulating hormone and estradiol levels test.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Evidence of a clinically significant (as judged by the Investigator) condition or abnormality (other than the indication being studied) that might compromise safety or the interpretation of trial efficacy or safety endpoints.
* Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
* A previous episode of treated tuberculosis less than 3 years ago.
* Clinically significant evidence of extrathoracic tuberculosis (miliary tuberculosis, abdominal tuberculosis, urogenital tuberculosis, osteoarthritic tuberculosis, tuberculosis meningitis), as judged by the Investigator.
* Corrected QT Interval > 450 milliseconds.
* History of allergy to any of the trial investigational product/s or related substances as confirmed by the clinical judgement of the Investigator.
* History of photosensitivity.
* Known or suspected, current or history of within the past 2 years, alcohol or drug abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the subject.
* HIV infected subjects: having a cluster of differentiation 4+ (CD4+) count <350 cells per microliter; or having received antiretroviral therapy medication within the last 90 days; or having received oral or intravenous antifungal medication within the last 90 days; or with an AIDS-defining opportunistic infection or malignancies (except pulmonary tuberculosis).
* Participated in other clinical studies with investigational agents within 8 weeks prior to the first dosing day in the current study.
* Subjects with diabetes (Type 1 or 2), point of care glycated hemoglobin above 6.5 millimoles per mole, or random glucose over 11.1 millimoles per liter will be excluded from cohorts undergoing FDGPET/CT. Subjects not undergoing FDG-PET/CT will be excluded if they have unstable diabetes or insulin dependency.
* Treatment received with any drug active against MTB (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole), or with immunosuppressive medications such as tumor necrosis factor -alpha inhibitors or systemic or inhaled corticosteroids, within 2 weeks prior to screening.
* Subjects with the following abnormal laboratory values at screening as defined by the enhanced Common Terminology Criteria for Adverse Events toxicity table: creatinine grade 2 or greater (>1.5 times upper limit of normal [ULN]); hemoglobin <10.0 grams per deciliter; thrombocytopenia grade 2 or greater (under 50 times 10^9 cells per liter); serum potassium grade 2 or greater (<3.0 milliequivalents per liter); aspartate aminotransferase grade 3 (>=3.0 times ULN); alanine aminotransferase grade 3 (>=3.0 times ULN); activated partial thromboplastin time grade 3 (>=2.5 times ULN); international normalized ratio grade 3 (>=2.5 times ULN); total white cell count grade 3 (<2.0 times 10^9 cells per liter).
* Subjects who are selected to undergo FDG-PET/CT who have been estimated to have been exposed to ionizing radiation in excess of 10 millisievert above background over the previous three-year period as a result of occupational exposure to radiation or as a result of research studies. This will be judged through clinical history taking.
* Women who are susceptible to heavy periods or heavy vaginal bleeding or spotting will be excluded in order to minimize blood loss and avoid confounding effects on the interpretation of hematology parameters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Diacon AH, Barry CE 3rd, Carlton A, Chen RY, Davies M, de Jager V, Fletcher K, Koh GCKW, Kontsevaya I, Heyckendorf J, Lange C, Reimann M, Penman SL, Scott R, Maher-Edwards G, Tiberi S, Vlasakakis G, Upton CM, Aguirre DB. A first-in-class leucyl-tRNA synthetase inhibitor, ganfeborole, for rifampicin-susceptible tuberculosis: a phase 2a open-label, randomized trial. Nat Med. 2024 Mar;30(3):896-904. doi: 10.1038/s41591-024-02829-7. Epub 2024 Feb 16. PMID 38365949
- [Derived] Volynets GP, Usenko MO, Gudzera OI, Starosyla SA, Balanda AO, Syniugin AR, Gorbatiuk OB, Prykhod'ko AO, Bdzhola VG, Yarmoluk SM, Tukalo MA. Identification of dual-targeted Mycobacterium tuberculosis aminoacyl-tRNA synthetase inhibitors using machine learning. Future Med Chem. 2022 Sep;14(17):1223-1237. doi: 10.4155/fmc-2022-0085. Epub 2022 Jul 25. PMID 35876255

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label trial to investigate the early bactericidal activity, safety and tolerability of GSK3036656 in participants with drug-sensitive pulmonary tuberculosis. Participants received Rifafour e-275 as a standard-of-care or GSK3036656. Rifafour e-275 is a registered trademark of Sanofi-Aventis company.
Pre-assignment Details: A total of 76 participants were enrolled (Enrolled Population consisted of all participants who passed screening and entered the study) in this study.
Groups:
- Rifafour e-275: All participants received a standard-of-care therapy ( rifafour e-275) tablet, orally, once daily from Day 1 to Day 14. Participants received the standard treatment for tuberculosis (i.e. rifafour e-275 or equivalent generic alternative) once the study treatment (Day 1 to Day 14) was completed.
- GSK3036656 1 mg: Participants received a loading dose of GSK3036656 3 milligram (mg), capsule, orally on Day 1, followed by maintenance dose of GSK3036656 1 mg, orally, once daily from Day 2 to Day 14.
- GSK3036656 5 mg: Participants received a loading dose of GSK3036656 15 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 5 mg, orally, once daily from Day 2 to Day 14.
- GSK3036656 15 mg: Participants received a loading dose of GSK3036656 30 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 15 mg, orally, once daily from Day 2 to Day 14.
- GSK3036656 30 mg: Participants received a loading dose of GSK3036656 75 mg, capsule, orally on Day 1, followed by maintenance dose of GSK3036656 30 mg, orally, once daily from Day 2 to Day 14.
Period: Overall Study
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Started | 18 | 9 | 17 | 16 | 16
Safety Population Consisted of All Randomized Participants Who Received at Least 1 Dose of Treatment | 18 | 9 | 17 | 16 | 15
Completed | 18 | 8 | 15 | 15 | 13
Not Completed | 0 | 1 | 2 | 1 | 3
Not completed — Investigator discretion | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 2
Not completed — Randomized, but did not receive treatment | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg | Total
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15 | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (10.20) | 37.8 (8.38) | 38.1 (10.33) | 39.8 (12.33) | 38.5 (9.82) | 38.2 (10.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 18 | 9 | 17 | 16 | 15 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 18 | 9 | 17 | 16 | 15 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in log10 Colony Forming Units (CFU) Per (/) Milliliter (mL) of Direct Respiratory Sputum Samples From Baseline to Day 14
Description: The Early Bactericidal Activity was determined by change in log10CFU/mL of sputum over the period Baseline to Day 14. Log(CFU) was calculated as: Log(CFU/mL)=log10(mean[Total count 1:Total Count 2]*2*5*10^Dilution); where total counts 1 and 2 were bacterial counts from plates 1 and 2 respectively; *2 represents the 1:1 dilution of the original specimen and *5 represents the 0.2 mL (200 microliter) inoculation of the specimen; Dilution is the dilution factor for that plate. Baseline (Day 0) was defined as the mean of Day -2 and Day -1; if data was available at only one of these timepoints then that value was used as Baseline.
Time Frame: Baseline and up to Day 14
Population: Efficacy Population consisted of participants in the safety population who provided at least two evaluable overnight sputum samples.
Measure: Mean (Standard Error); unit: Log10CFU/mL
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
Log10CFU/mL | -0.199 (0.0130) | -0.017 (0.0182) | -0.092 (0.0136) | -0.092 (0.0142) | -0.138 (0.0147)

2. Secondary Outcome: Change in log10 CFU/mL of Direct Respiratory Sputum Samples From Baseline to Day 2
Description: The Early Bactericidal Activity was determined by change in log10CFU per mL of sputum over the period Baseline to Day 2. Log(CFU) was calculated as: Log(CFU/mL)=log10(mean[Total count 1:Total Count 2]*2*5*10^Dilution); where total counts 1 and 2 were bacterial counts from plates 1 and 2 respectively; *2 represents the 1:1 dilution of the original specimen and *5 represents the 0.2 mL (200 microliter) inoculation of the specimen; Dilution is the dilution factor for that plate. Baseline (Day 0) was defined as the mean of Day -2 and Day -1; if data was available at only one of these timepoints then that value was used as Baseline.
Time Frame: Baseline and up to Day 2
Population: Efficacy Population consisted of participants in the safety population who provided at least two evaluable overnight sputum samples. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Error); unit: log10CFU/mL
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 17 | 9 | 17 | 16 | 15
log10CFU/mL | -0.598 (0.0801) | 0.250 (0.1077) | -0.153 (0.0801) | -0.055 (0.0832) | -0.040 (0.0855)

3. Secondary Outcome: Change in log10 CFU Per mL of Direct Respiratory Sputum Samples From Day 2 to Day 14
Description: The Early Bactericidal Activity was determined by change in log10CFU per mL of sputum over the period Day 2 to Day 14. Log(CFU) was calculated as: Log(CFU/mL)=log10(mean[Total count 1:Total Count 2]*2*5*10^Dilution); where total counts 1 and 2 were bacterial counts from plates 1 and 2 respectively; *2 represents the 1:1 dilution of the original specimen and *5 represents the 0.2 mL (200 microliter) inoculation of the specimen; Dilution is the dilution factor for that plate.
Time Frame: Day 2 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log10CFU/mL
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 17 | 9 | 16 | 16 | 14
log10CFU/mL | -0.162 (0.0169) | -0.037 (0.0233) | -0.080 (0.0173) | -0.086 (0.0181) | -0.129 (0.0192)

4. Secondary Outcome: Change in log10 Time to Sputum Culture Positivity (TTP) From Baseline to Day 14
Description: The Early Bactericidal Activity was determined by change in TTP per mL sputum over the period Baseline to Day 14. The TTP was measured in the Mycobacterial Growth Indicator Tube (MGIT) automated liquid culture system of time to positivity of Mycobacterium tuberculosis from an overnight sputum collection. Time to sputum-culture positivity was the time between sample inoculation and detection of mycobacterial growth in the mycobacterium growth indicator tube. Baseline (Day 0) was defined as the mean of Day -2 and Day -1; if data was available at only one of these timepoints then that value was used as Baseline.
Time Frame: Baseline and up to Day 14
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10hours
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
log10hours | 0.025 (0.0010) | 0.000 (0.0015) | 0.015 (0.0011) | 0.021 (0.0012) | 0.022 (0.0013)

5. Secondary Outcome: Change in log10 TTP From Baseline to Day 2
Description: The Early Bactericidal Activity was determined by change in TTP per mL sputum over the period Baseline to Day 2. The TTP was measured in the MGIT automated liquid culture system of time to positivity of Mycobacterium tuberculosis from an overnight sputum collection. Time to sputum-culture positivity was the time between sample inoculation and detection of mycobacterial growth in the mycobacterium growth indicator tube. Baseline (Day 0) was defined as the mean of Day -2 and Day -1; if data was available at only one of these timepoints then that value was used as Baseline.
Time Frame: Baseline and up to Day 2
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10hours
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
log10hours | 0.105 (0.0068) | -0.003 (0.0096) | 0.021 (0.0071) | 0.032 (0.0072) | 0.066 (0.0074)

6. Secondary Outcome: Change in log10 TTP From Day 2 to Day 14
Description: The Early Bactericidal Activity was determined by change in TTP per mL sputum over the period Day 2 to Day 14. The TTP was measured in the MGIT automated liquid culture system of time to positivity of Mycobacterium tuberculosis from an overnight sputum collection. Time to sputum-culture positivity was the time between sample inoculation and detection of mycobacterial growth in the mycobacterium growth indicator tube.
Time Frame: Day 2 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Error); unit: log10hours
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 16 | 16 | 15
log10hours | 0.017 (0.0011) | 0.001 (0.0016) | 0.013 (0.0012) | 0.017 (0.0012) | 0.016 (0.0013)

7. Secondary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve From Time Zero to Last Time of Quantifiable Concentration (AUC[0-t]) Following Once Daily Dosing of GSK3036656
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3036656.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: PK Population consisted of participants in the safety population who received at least one dose of GSK3036656 and had at least one evaluable PK sample. Only those participants with data available at specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 8 | 14 | 14 | 13
Hours*nanogram per milliliter | 281.8 (25.7) | 1495.6 (12.5) | 4493.8 (12.5) | 11505.6 (17.9)

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Zero to 24 Hours (AUC[0-24]) Following Once Daily Dosing of GSK3036656
Description: Blood samples were collected at indicated time points for PK analysis of GSK3036656.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 8 | 14 | 14 | 13
Hours*nanogram per milliliter | 282.1 (25.8) | 1497.1 (12.4) | 4493.9 (12.5) | 11540.0 (17.8)

9. Secondary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) Following Once Daily Dosing of GSK3036656
Description: Blood samples were collected at indicated time points for PK analysis of GSK3036656.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 8 | 14 | 14 | 13
Nanogram per milliliter | 16.93 (23.7) | 94.60 (24.7) | 291.41 (18.9) | 705.24 (20.2)

10. Secondary Outcome: Time to Reach Cmax (Tmax) Following Once Daily Dosing of GSK3036656
Description: Blood samples were collected at indicated time points for PK analysis of GSK3036656.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose on Day 14
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 8 | 14 | 14 | 13
Hours | 1.500 [0.50 to 6.00] | 2.492 [0.50 to 4.00] | 1.000 [0.50 to 4.00] | 2.000 [0.50 to 8.00]

11. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Adverse events which were not Serious Adverse Events were considered as Non-Serious adverse events.
Time Frame: Up to Day 28 (follow-up visit)
Population: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
Participants
  Non-SAEs | 14 | 7 | 14 | 15 | 9
  SAEs1 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, total neutrophils, and platelet count. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: Safety Population consisted of all randomized participants who received at least one dose of study treatment. Only those participants with data available at specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
10^9 cells per liter
  Basophils | -0.006 (0.0281) | -0.009 (0.0242) | -0.018 (0.0248) | -0.003 (0.0263) | -0.005 (0.0267)
  Eosinophils | 0.086 (0.1383) | 0.075 (0.1135) | 0.088 (0.1239) | 0.072 (0.0880) | 0.057 (0.0642)
  Lymphocytes | 0.051 (0.3024) | -0.066 (0.3066) | 0.157 (0.4010) | 0.099 (0.5175) | 0.136 (0.3861)
  Monocytes | -0.073 (0.3236) | -0.156 (0.1467) | -0.125 (0.1376) | -0.301 (0.3647) | -0.242 (0.2225)
  Total neutrophils | -0.940 (1.9563) | -0.509 (0.9609) | -0.613 (1.4654) | -1.633 (1.6475) | -0.949 (1.2011)
  Platelet count: number analyzed (Participants) | 17 | 8 | 15 | 15 | 13
  Platelet count | -59.6 (105.19) | -35.0 (83.00) | -93.6 (81.05) | -7.3 (81.33) | -78.6 (43.53)

13. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Grams per liter | -3.4 (9.15) | -2.9 (6.64) | 0.0 (7.32) | 1.7 (9.21) | -4.6 (14.99)

14. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Proportion of red blood cells in blood | -0.012 (0.0308) | -0.008 (0.0225) | 0.003 (0.0247) | 0.007 (0.0277) | -0.018 (0.0454)

15. Secondary Outcome: Change From Baseline in Hematology Parameter: Red Blood Cells Count
Description: Blood samples were collected to analyze the hematology parameter: red blood cells count. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
10^12 cells per liter | -0.130 (0.3067) | -0.091 (0.2776) | 0.016 (0.2753) | 0.059 (0.2875) | -0.216 (0.6590)

16. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: mean corpuscular volume. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Femtoliter | 0.2 (1.92) | -0.3 (0.89) | 0.1 (1.36) | 0.5 (0.92) | 0.0 (1.35)

17. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: mean corpuscle hemoglobin. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Picograms | 0.2 (0.65) | -0.1 (0.64) | -0.1 (0.64) | 0.1 (0.70) | 0.3 (0.75)

18. Secondary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes
Description: Blood samples were collected to analyze the hematology parameter: reticulocytes. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Percentage of reticulocytes | 0.0045 (0.00568) | 0.0035 (0.00245) | 0.0041 (0.00255) | 0.0055 (0.00374) | 0.0025 (0.00456)

19. Secondary Outcome: Change From Baseline in Chemistry Parameters: Glucose, Calcium, Chloride, Potassium, Sodium, Blood Urea Nitrogen
Description: Blood samples were collected to analyze the chemistry parameters: glucose, calcium, chloride, potassium, sodium, and blood urea nitrogen. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Millimoles per liter
  Glucose | -0.29 (0.734) | 0.05 (0.809) | 0.17 (1.047) | -0.30 (0.902) | -0.86 (1.477)
  Calcium | 0.021 (0.0814) | -0.018 (0.1007) | -0.034 (0.0672) | 0.005 (0.0633) | -0.024 (0.0860)
  Chloride | 1.1 (2.14) | 1.0 (1.69) | 1.6 (2.59) | 2.3 (2.25) | 2.3 (3.79)
  Potassium | -0.39 (0.398) | -0.79 (0.925) | -0.47 (0.403) | -0.15 (0.521) | -0.28 (0.521)
  Sodium | 0.4 (2.33) | 1.0 (1.60) | 0.7 (2.55) | 2.1 (3.49) | 0.5 (3.10)
  Blood urea nitrogen | -0.054 (0.3207) | -0.169 (0.5493) | 0.125 (0.3074) | 0.145 (0.2860) | 0.042 (0.3198)

20. Secondary Outcome: Change From Baseline in Chemistry Parameters: Lactate Dehydrogenase (LDH), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT)
Description: Blood samples were collected to analyze the chemistry parameters: LDH, ALT, ALP, AST and GGT. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
International units per liter
  LDH | -56.3 (57.81) | -52.8 (72.99) | -18.3 (36.22) | -26.5 (57.92) | -8.5 (73.83)
  ALT | -20.6 (35.79) | -37.0 (62.35) | -8.1 (18.22) | -11.0 (18.60) | 5.9 (20.77)
  ALP | -3.1 (21.22) | -34.1 (61.88) | -16.8 (32.52) | -4.0 (70.73) | -7.5 (13.06)
  AST | -13.7 (22.27) | -12.9 (13.94) | -5.6 (9.86) | -8.4 (13.47) | 2.2 (8.74)
  GGT | -3.9 (22.20) | -51.0 (76.64) | -14.9 (28.18) | -16.4 (30.83) | -5.2 (23.23)

21. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine, Indirect Bilirubin, Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: creatinine, indirect bilirubin, direct bilirubin and total bilirubin. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Micromoles per liter
  Creatinine | 0.6 (6.09) | 2.8 (4.74) | 3.1 (9.13) | 1.5 (6.24) | 0.6 (5.08)
  Indirect bilirubin: number analyzed (Participants) | 15 | 7 | 15 | 15 | 13
  Indirect bilirubin | -1.2 (1.08) | -0.9 (1.07) | -0.1 (1.51) | -1.1 (1.71) | 0.3 (1.03)
  Direct bilirubin | -0.6 (0.70) | -0.5 (1.07) | 0.0 (0.76) | -0.7 (0.90) | -0.7 (1.38)
  Total bilirubin | -1.5 (1.34) | -1.1 (1.81) | -0.1 (1.51) | -1.7 (2.05) | 0.0 (1.58)

22. Secondary Outcome: Change From Baseline in Chemistry Parameter: Total Protein
Description: Blood samples were collected to analyze the chemistry parameter: total protein. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Grams per liter | -1.7 (3.72) | -1.0 (6.46) | -1.3 (4.73) | 2.2 (6.73) | -4.2 (5.83)

23. Secondary Outcome: Number of Participants With Worst-Case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method
Description: Urine samples were collected to assess urine occult blood and urine protein. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as no change/decreased and increase to abnormal for urine occult blood and protein indicating proportional concentrations in the urine sample. 'No change/decreased' means no change from Baseline or a value less than the Baseline value. 'Increase to abnormal' means an increase from the Baseline value that is considered as an abnormal value. Baseline value is the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline (Day 1, Pre-dose) and up to Day 28 (follow-up visit)
Population: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
Participants
  Occult blood: No change/decrease | 15 | 9 | 16 | 14 | 9
  Occult blood: Increase to abnormal | 3 | 0 | 1 | 2 | 6
  Protein: No change/decrease | 8 | 5 | 9 | 10 | 9
  Protein: Increase to abnormal | 10 | 4 | 8 | 6 | 6

24. Secondary Outcome: Number of Participants With Worst Case Vital Sign Results by Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Vital signs were measured in a semi-supine or supine position after 5 minutes rest. The PCI range for vital signs were: systolic blood pressure (SBP) (lower: <85 and upper: >160 milliliter of mercury [mmHg]); diastolic blood pressure (DBP) (lower: <45 and upper: >100 mmHg); heart rate (lower: <40 and upper: >110 beats per minute [bpm]); respiratory rate (lower: 10 and upper: 28 breaths per minutes) and temperature (lower: <35 and upper: >37.9 degrees Celsius). Participants were counted in the worst-case category that their value changed to (low, within range or no change, or high), unless there was no change in their category. Participants whose value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To w/in Range or No Change category". Participants were counted twice if the participant had values that changed "To Low" and "To High".
Time Frame: Up to Day 28 (follow-up visit)
Population: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 17 | 16 | 15
Participants
  SBP: To low | 1 | 1 | 0 | 1 | 0
  SBP: To within Range or No Change | 17 | 8 | 17 | 15 | 15
  SBP: To High | 0 | 0 | 0 | 0 | 0
  DBP: To low | 1 | 1 | 1 | 0 | 0
  DBP: To within Range or No Change | 16 | 7 | 16 | 16 | 15
  DBP: To High | 1 | 1 | 0 | 0 | 0
  Heart rate: To low | 0 | 0 | 0 | 0 | 0
  Heart rate: To within Range or No Change | 16 | 6 | 15 | 15 | 15
  Heart rate: To High | 2 | 3 | 2 | 1 | 0
  Respiratory rate: To low | 0 | 0 | 0 | 0 | 0
  Respiratory rate: To within Range or No Change | 18 | 9 | 17 | 13 | 15
  Respiratory rate: To High | 0 | 0 | 0 | 3 | 0
  Temperature: To low | 0 | 0 | 0 | 1 | 0
  Temperature: To within Range or No Change | 17 | 7 | 16 | 14 | 15
  Temperature: To High | 1 | 2 | 1 | 1 | 0

25. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, uncorrected QT and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal laboratory findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with abnormal clinically significant ECG findings for worst case post-Baseline has been presented.
Time Frame: Up to Day 28 (follow-up visit)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 9 | 15 | 16 | 15
Participants
  Abnormal, not clinically significant | 13 | 5 | 12 | 12 | 10
  Abnormal - clinically significant | 0 | 0 | 0 | 1 | 0

26. Secondary Outcome: Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF)
Description: Twelve-lead ECGs were obtained to QTcF Interval and measured QT duration corrected for heart rate by Fridericia's formula interval. Baseline value was the latest assessment prior to Day 1 dose with a non-missing value, including those from unscheduled visits and the mean of the triplicate measurements at any given time point was used as the value for that time point. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit (Day 14) value.
Time Frame: Baseline (Day 1, Pre-dose) and at Day 14
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
Number analyzed (Participants) | 18 | 8 | 15 | 15 | 13
Milliseconds | 6.4 (13.64) | 11.3 (14.40) | -1.8 (20.48) | 9.5 (14.91) | 4.0 (16.76)

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected up to Day 28 (follow-up visit)
Description: Safety Population consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Rifafour e-275 | GSK3036656 1 mg | GSK3036656 5 mg | GSK3036656 15 mg | GSK3036656 30 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/9 | 0/17 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/9 | 0/17 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 14/18 | 7/9 | 14/17 | 15/16 | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifafour e-275 (N=18) | GSK3036656 1 mg (N=9) | GSK3036656 5 mg (N=17) | GSK3036656 15 mg (N=16) | GSK3036656 30 mg (N=15)
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Noninfective myringitis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03557281/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT03557281/SAP_001.pdf